CLINICAL TRIAL: NCT06282432
Title: Long-Term Follow-Up (LTFU) for Gene Therapy of Leukocyte Adhesion Deficiency-I (LAD-I) Phase I/II Clinical Study to Evaluate the Safety and Efficacy of the Infusion of Autologous Hematopoietic Stem Cells Transduced With a Lentiviral Vector Encoding the ITGB2 Gene
Brief Title: Long-Term Follow-Up (LTFU) for Gene Therapy of Leukocyte Adhesion Deficiency-I (LAD-I)
Status: Active, not recruiting | Type: Observational
Sponsor: Rocket Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RP-L201-0121-LTFU
Record Dates: First submitted 2023-11-13; First posted 2024-02-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Leukocyte Adhesion Deficiency
Keywords: LAD-I; LAD
MeSH Terms: conditions — Leukocyte adhesion deficiency type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human Tissue (including blood and bone marrow)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects that received RP-L201 on the RP-L201-0318 Parent Study: Subjects that received RP-L201 on the RP-L201-0318 Parent Study and either completed the study or discontinued early.

SUMMARY:
This Long-Term Follow-Up (LTFU) for Gene Therapy of Leukocyte Adhesion Deficiency-I (LAD-I) is a continuation of a Phase 1/2 clinical study to evaluate the safety and efficacy of the infusion of autologous hematopoietic stem cells transduced with a lentiviral vector encoding the ITGB2 gene

DETAILED DESCRIPTION:
Following the end of participation in Study RP-L201-0318, patients will be offered enrollment into this LTFU protocol. Patients will be followed for up to 15 years following the RP-L201 infusion in the parent study, until the patient dies, withdraws consent, or is lost to follow-up (whichever occurs first).

For all follow-up visits, remote evaluation facilitated by local health care providers (with blood sample shipment to relevant laboratory facilities) is permitted; however, annual visits to the study center are required during initial 3 years post- RP-L201 infusion. Visits where a bone marrow sample is being collected are required to be performed at the study center for the duration of the study. Peripheral Blood samples and bone marrow samples will be archived and tested when clinically or scientifically indicated, as in the event of development of a second malignancy.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in the Phase I/II Study RP-L201-0318.
2. Received an autologous infusion of CD34+ hematopoietic stem cells modified with a lentiviral vector containing the ITGB2 gene, encoding for the human CD18 receptor in the parent Study RP-L201-0318.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Provided written informed consent and, as applicable, assent to participate in the current study.

Exclusion Criteria:

There are no criteria for exclusion in this study.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects that have been treated with RP-L201 on the RP-L201-0318 study.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2036-10-04 (Estimated); Study Completion 2036-10-04 (Estimated)

PRIMARY OUTCOMES:
Hematopoietic stem cell transplant (HSCT) free survival | 15 years
  Survival without allogeneic-HSCT.

SECONDARY OUTCOMES:
Incidence of hospitalizations | 15 years
  Incidence of infection-related hospitalizations.
Incidence of significant infections | 15 years
  Incidence of infections requiring hospitalization or intravenous antimicrobials.
Resolution of LAD-I-related skin rash | 15 years
  Partial or complete resolution of LAD-I skin rash evident by photographical images.
Resolution of LAD-I-related periodontal abnormalities | 15 years
  Partial or complete resolution of LAD-I periodontal abnormalities evident by photographical images.
Event free survival | 15 years
  Survival in the absence of graft failure and graft versus host disease.
Overall Survival | 15 years
  Survival in the absence of death from any cause
Long-term genetic correction in peripheral blood mononuclear cells (PBMCs) | 15 years
  Persistence of transgene in PB cells as demonstrated by vector copy number (VCN) of at least 0.1 in PBMCs.
Long-term genetic correction in PB CD15+ granulocytes | 15 years
  Persistence of transgene in PB cells as demonstrated by VCN of at least 0.1 in PB CD15+ granulocytes.
Long-term CD18 neutrophil expression by flow cytometry | 15 Years
  Persistence of CD18 neutrophil expression defined by PB neutrophil CD18 expression to at least 10% of normal.
Long-term CD11 neutrophil expression by flow cytometry | 15 Years
  Persistence of CD11 a/b neutrophil co-expression
Improvement or resolution of LAD-I related neutrophilia | 15 Years
  Improvement of LAD-I related neutrophilia based off neutrophils within age-appropriate normal ranges.
Improvement or resolution of LAD-I-related leukocytosis. | 15 Years
  Improvement of LAD-I related leukocytosis based off leukocytes within age-appropriate normal ranges.
Incidence of Investigational Product (IP) related serious adverse events (SAEs) | 15 Years
  Incidence of SAEs related to the IP measured by CTCAE (Common Terminology Criteria for Adverse Events) for V5.0 grading scale.
Incidence of hematologic malignancy | 15 Years
  Incidence of hematologic malignancy related to prior gene therapy or gene-therapy associated medications.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Kohn, MD, Principal Investigator — University of California, Los Angeles; Claire Booth, MBBS, PhD, MSc, Principal Investigator — University College London Great Ormond Street Institute of Child Health; Julian Sevilla, MD, PhD, Principal Investigator — Hospital Infantil Universitario Niño Jesús
Locations (3):
- University of California, Los Angeles (UCLA), Los Angeles, California, United States
- Hospital Infantil Universitario Niño Jesús, Madrid, Spain
- University College London Great Ormond Street Institute of Child Health (GOSH), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Booth C, Sevilla J, Almarza E, Kuo CY, Zubicaray J, Terrazas D, O'Toole G, Chitty-Lopez M, Choi G, Nicoletti E, Long-Boyle J, Fernandes A, Chetty K, De Oliveira S, Banuelos C, Xu-Bayford J, Bastone AL, John-Neek P, Jackson C, Moore TB, Gilmour K, Schambach A, Rothe M, Kasbekar S, Rao GR, Patel K, Shah G, Thrasher AJ, Bueren JA, Schwartz JD, Kohn DB. Lentiviral Gene Therapy for Severe Leukocyte Adhesion Deficiency Type 1. N Engl J Med. 2025 May 1;392(17):1698-1709. doi: 10.1056/NEJMoa2407376. PMID 40305711